CLINICAL TRIAL: NCT00680186
Title: A Phase III, Randomised, Double Blind, Parallel-group Study of the Efficacy and Safety of Oral Dabigatran Etexilate (150 mg Bid) Compared to Warfarin (INR 2.0-3.0) for 6 Month Treatment of Acute Symptomatic Venous Thromboembolism, Following Initial Treatment (5-10 Days) With a Parenteral Anticoagulant Approved for This Indication
Brief Title: Phase III Study Testing Efficacy & Safety of Oral Dabigatran Etexilate vs Warfarin for 6 m Treatment for Acute Symp Venous Thromboembolism (VTE)
Acronym: RE-COVER II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1160.46; 2007-002631-86 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Results first posted 2012-06-14 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2013-12

CONDITIONS: Thromboembolism
MeSH Terms: conditions — Thromboembolism | interventions — Warfarin; Dabigatran

ARMS (2):
- Dabigatran etexilate (150mg bid) (Experimental): Patients will receive 1 capsule containing 150 mg dabigatran etexilate/matching placebo twice daily
  Interventions: Drug: Dabigatran etexilate
- Warfarin (INR 2.0-3.0) (Active Comparator): Patients will receive tablets PRN warfarin/matching placebo to maintain a target INR of 2.0-3.0
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — PRN (to maintain a target INR of 2.0-3.0)
  Arms: Warfarin (INR 2.0-3.0)
Drug: Dabigatran etexilate — 150mg bid
  Arms: Dabigatran etexilate (150mg bid)

SUMMARY:
The general aim of this study is to determine the comparative safety and efficacy of dabigatran etexilate 150 mg bid administered orally and warfarin Pro re nata (As needed/PRN) to maintain an International Normalised Ratio (INR) of 2.0-3.0 for 6 month treatment of acute symptomatic VTE.

The primary objective is to investigate the efficacy of dabigatran compared to warfarin during the 6 month treatment period. The investigation of other selected efficacy aspects and safety are regarded as secondary objective of this trial.

ELIGIBILITY:
Inclusion criteria:

* Acute symptomatic uni- or bilateral Deep Vein Thrombosis (DVT) of the leg involving proximal veins, and/or Pulmonary Embolism (PE)
* Male or female, being 18 years of age or older
* Written informed consent for study participation

Exclusion criteria:

* Persistent symptoms of VTE
* PE requiring urgent intervention
* Use of vena cava filter
* Contraindications to anticoagulant therapy
* Allergy to study medications
* Elevated Aspartate-aminotransferase (AST) or Alanine-aminotransferase (ALT) > 3x Upper Limit of Normal (ULN) or known liver disease expected to have an impact on survival
* Severe renal impairment
* Patients considered unsuitable for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2589 (Actual)
Dates: Start 2008-04; Primary Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (220):
- United States (10):
  - 1160.46.01073 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 1160.46.01044 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1160.46.01068 Boehringer Ingelheim Investigational Site, Normal, Illinois
  - 1160.46.01071 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 1160.46.01060 Boehringer Ingelheim Investigational Site, Stony Brook, New York
  - 1160.46.01061 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1160.46.01059 Boehringer Ingelheim Investigational Site, Bend, Oregon
  - 1160.46.01063 Boehringer Ingelheim Investigational Site, Corvallis, Oregon
  - 1160.46.01055 Boehringer Ingelheim Investigational Site, Summerville, South Carolina
  - 1160.46.01062 Boehringer Ingelheim Investigational Site, Bellevue, Washington
- Australia (5):
  - 1160.46.61007 Boehringer Ingelheim Investigational Site, Concord, New South Wales
  - 1160.46.61003 Boehringer Ingelheim Investigational Site, Box Hill, Victoria
  - 1160.46.61001 Boehringer Ingelheim Investigational Site, Clayton, Victoria
  - 1160.46.61006 Boehringer Ingelheim Investigational Site, Windsor, Victoria
  - 1160.46.61005 Boehringer Ingelheim Investigational Site, Perth, Western Australia
- Brazil (9):
  - 1160.46.55010 Boehringer Ingelheim Investigational Site, Brasília
  - 1160.46.55007 Boehringer Ingelheim Investigational Site, Campinas
  - 1160.46.55014 Boehringer Ingelheim Investigational Site, Curitiba
  - 1160.46.55017 Boehringer Ingelheim Investigational Site, Curitiba
  - 1160.46.55019 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1160.46.55021 Boehringer Ingelheim Investigational Site, Recife
  - 1160.46.55016 Boehringer Ingelheim Investigational Site, Rio de Janeiro - RJ
  - 1160.46.55018 Boehringer Ingelheim Investigational Site, São Bernardo do Campo
  - 1160.46.55020 Boehringer Ingelheim Investigational Site, São Paulo
- Bulgaria (4):
  - 1160.46.35901 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.46.35903 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.46.35906 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.46.35905 Boehringer Ingelheim Investigational Site, Varna
- Canada (15):
  - 1160.46.02006 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1160.46.02013 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1160.46.02021 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 1160.46.02004 Boehringer Ingelheim Investigational Site, Saint John, New Brunswick
  - 1160.46.02001 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 1160.46.02002 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.46.02005 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.46.02010 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.46.02015 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1160.46.02019 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1160.46.02008 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.46.02009 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.46.02014 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.46.02017 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.46.02020 Boehringer Ingelheim Investigational Site, Québec, Quebec
- China (16):
  - 1160.46.86001 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.46.86002 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.46.86019 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.46.86014 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1160.46.86015 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1160.46.86016 Boehringer Ingelheim Investigational Site, Hangzhou
  - 1160.46.86003 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.46.86004 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.46.86005 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.46.86011 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.46.86007 Boehringer Ingelheim Investigational Site, Shenyang
  - 1160.46.86017 Boehringer Ingelheim Investigational Site, Shijiazhuang
  - 1160.46.86018 Boehringer Ingelheim Investigational Site, Shijiazhuang
  - 1160.46.86021 Boehringer Ingelheim Investigational Site, Taiyuan
  - 1160.46.86006 Boehringer Ingelheim Investigational Site, Tianjin
  - 1160.46.86020 Boehringer Ingelheim Investigational Site, Yinchuan
- Czechia (11):
  - 1160.46.42001 Boehringer Ingelheim Investigational Site, Brno
  - 1160.46.42002 Boehringer Ingelheim Investigational Site, Hradec Králové
  - 1160.46.42012 Boehringer Ingelheim Investigational Site, Liberec
  - 1160.46.42018 Boehringer Ingelheim Investigational Site, Litoměřice
  - 1160.46.42015 Boehringer Ingelheim Investigational Site, Nový Jičín
  - 1160.46.42005 Boehringer Ingelheim Investigational Site, Ostrava-Vitkovice
  - 1160.46.42017 Boehringer Ingelheim Investigational Site, Prague
  - 1160.46.42014 Boehringer Ingelheim Investigational Site, Tábor
  - 1160.46.42016 Boehringer Ingelheim Investigational Site, Teplice
  - 1160.46.42010 Boehringer Ingelheim Investigational Site, Ústí nad Labem
  - 1160.46.42007 Boehringer Ingelheim Investigational Site, Zlín
- Denmark (4):
  - 1160.46.45001 Boehringer Ingelheim Investigational Site, Aarhus C
  - 1160.46.45008 Boehringer Ingelheim Investigational Site, Esbjerg
  - 1160.46.45009 Boehringer Ingelheim Investigational Site, Holbæk
  - 1160.46.45004 Boehringer Ingelheim Investigational Site, København NV
- France (15):
  - 1160.46.3301A Boehringer Ingelheim Investigational Site, Brest
  - 1160.46.3301B Boehringer Ingelheim Investigational Site, Brest
  - 1160.46.3315A Boehringer Ingelheim Investigational Site, La Roche-sur-Yon
  - 1160.46.3315B Boehringer Ingelheim Investigational Site, La Roche-sur-Yon
  - 1160.46.3313A Boehringer Ingelheim Investigational Site, Nantes
  - 1160.46.3316A Boehringer Ingelheim Investigational Site, Pessac
  - 1160.46.3316B Boehringer Ingelheim Investigational Site, Pessac
  - 1160.46.3303C Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1160.46.3303D Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1160.46.3303E Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1160.46.3303F Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1160.46.3303G Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1160.46.3303H Boehringer Ingelheim Investigational Site, Saint-Etienne
  - 1160.46.3303A Boehringer Ingelheim Investigational Site, Saint-Priest-en-Jarez
  - 1160.46.3303B Boehringer Ingelheim Investigational Site, Saint-Priest-en-Jarez
- Hungary (3):
  - 1160.46.36002 Boehringer Ingelheim Investigational Site, Debrecen
  - 1160.46.36010 Boehringer Ingelheim Investigational Site, Székesfehérvár
  - 1160.46.36011 Boehringer Ingelheim Investigational Site, Szombathely
- India (14):
  - 1160.46.91006 Boehringer Ingelheim Investigational Site, Bangalore
  - 1160.46.91010 Boehringer Ingelheim Investigational Site, Bangalore
  - 1160.46.91002 Boehringer Ingelheim Investigational Site, Chennai
  - 1160.46.91007 Boehringer Ingelheim Investigational Site, Chennai
  - 1160.46.91012 Boehringer Ingelheim Investigational Site, Kolkata
  - 1160.46.91009 Boehringer Ingelheim Investigational Site, Ludhiana
  - 1160.46.91008 Boehringer Ingelheim Investigational Site, Nagpur
  - 1160.46.91005 Boehringer Ingelheim Investigational Site, New Delhi
  - 1160.46.91014 Boehringer Ingelheim Investigational Site, New Delhi
  - 1160.46.91001 Boehringer Ingelheim Investigational Site, Pune
  - 1160.46.91004 Boehringer Ingelheim Investigational Site, Pune
  - 1160.46.91011 Boehringer Ingelheim Investigational Site, Tamil Nadu
  - 1160.46.91013 Boehringer Ingelheim Investigational Site, Vadodara
  - 1160.46.91003 Boehringer Ingelheim Investigational Site, Vadodra
- Israel (11):
  - 1160.46.97202 Boehringer Ingelheim Investigational Site, Afula
  - 1160.46.97207 Boehringer Ingelheim Investigational Site, Ashkelon
  - 1160.46.97212 Boehringer Ingelheim Investigational Site, DN Lower Galillee
  - 1160.46.97211 Boehringer Ingelheim Investigational Site, Haifa
  - 1160.46.97203 Boehringer Ingelheim Investigational Site, Holon
  - 1160.46.97205 Boehringer Ingelheim Investigational Site, KfarSaba
  - 1160.46.97209 Boehringer Ingelheim Investigational Site, Nazareth
  - 1160.46.97206 Boehringer Ingelheim Investigational Site, Petah Tikva
  - 1160.46.97210 Boehringer Ingelheim Investigational Site, Tel Aviv
  - 1160.46.97204 Boehringer Ingelheim Investigational Site, Tel Hashomer, Ramat Gan
  - 1160.46.97201 Boehringer Ingelheim Investigational Site, Ẕerifin
- Italy (6):
  - 1160.46.39011 Boehringer Ingelheim Investigational Site, Catania
  - 1160.46.39015 Boehringer Ingelheim Investigational Site, Florence
  - 1160.46.39012 Boehringer Ingelheim Investigational Site, Palermo
  - 1160.46.39007 Boehringer Ingelheim Investigational Site, Reggio Emilia
  - 1160.46.39013 Boehringer Ingelheim Investigational Site, Verona
  - 1160.46.39005 Boehringer Ingelheim Investigational Site, Vittorio Veneto (TV)
- Malaysia (4):
  - 1160.46.60001 Boehringer Ingelheim Investigational Site, Kelantan Kota Bahru
  - 1160.46.60004 Boehringer Ingelheim Investigational Site, Kuala Pahang
  - 1160.46.60002 Boehringer Ingelheim Investigational Site, Kuala Selangor
  - 1160.46.60003 Boehringer Ingelheim Investigational Site, Malacca
- Netherlands (8):
  - 1160.46.31010 Boehringer Ingelheim Investigational Site, 's-Hertogenbosch
  - 1160.46.31017 Boehringer Ingelheim Investigational Site, Alkmaar
  - 1160.46.31001 Boehringer Ingelheim Investigational Site, Amersfoort
  - 1160.46.31013 Boehringer Ingelheim Investigational Site, Eindhoven
  - 1160.46.31014 Boehringer Ingelheim Investigational Site, Heerlen
  - 1160.46.31002 Boehringer Ingelheim Investigational Site, Nieuwegein
  - 1160.46.31004 Boehringer Ingelheim Investigational Site, Rotterdam
  - 1160.46.31015 Boehringer Ingelheim Investigational Site, Zwolle
- New Zealand (4):
  - 1160.46.64004 Boehringer Ingelheim Investigational Site, Christchurch
  - 1160.46.64003 Boehringer Ingelheim Investigational Site, Grafton Auckland
  - 1160.46.64002 Boehringer Ingelheim Investigational Site, Otahuhu Auckland
  - 1160.46.64001 Boehringer Ingelheim Investigational Site, Takapuna Auckland
- Norway (2):
  - 1160.46.47001 Boehringer Ingelheim Investigational Site, Oslo
  - 1160.46.47005 Boehringer Ingelheim Investigational Site, Trondheim
- Philippines (4):
  - 1160.46.63005 Boehringer Ingelheim Investigational Site, City of Muntinlupa
  - 1160.46.63001 Boehringer Ingelheim Investigational Site, Manila
  - 1160.46.63003 Boehringer Ingelheim Investigational Site, Quezon City
  - 1160.46.63004 Boehringer Ingelheim Investigational Site, Quezon City
- Poland (5):
  - 1160.46.48004 Boehringer Ingelheim Investigational Site, Kielce
  - 1160.46.48001 Boehringer Ingelheim Investigational Site, Krakow
  - 1160.46.48005 Boehringer Ingelheim Investigational Site, Krakow
  - 1160.46.48003 Boehringer Ingelheim Investigational Site, Poznan
  - 1160.46.48006 Boehringer Ingelheim Investigational Site, Warsaw
- Russia (9):
  - 1160.46.07021 Boehringer Ingelheim Investigational Site, Chelyabinsk
  - 1160.46.07016 Boehringer Ingelheim Investigational Site, Krasnodar
  - 1160.46.07004 Boehringer Ingelheim Investigational Site, Kursk
  - 1160.46.07009 Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - 1160.46.07024 Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - 1160.46.07014 Boehringer Ingelheim Investigational Site, Ufa
  - 1160.46.07005 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 1160.46.07006 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 1160.46.07007 Boehringer Ingelheim Investigational Site, Yekaterinburg
- Singapore (3):
  - 1160.46.65001 Boehringer Ingelheim Investigational Site, Singapore
  - 1160.46.65002 Boehringer Ingelheim Investigational Site, Singapore
  - 1160.46.65003 Boehringer Ingelheim Investigational Site, Singapore
- Slovakia (4):
  - 1160.46.42107 Boehringer Ingelheim Investigational Site, Banská Bystrica
  - 1160.46.42106 Boehringer Ingelheim Investigational Site, Lučenec
  - 1160.46.42102 Boehringer Ingelheim Investigational Site, Nitra
  - 1160.46.42103 Boehringer Ingelheim Investigational Site, Nové Zámky
- South Africa (8):
  - 1160.46.27001 Boehringer Ingelheim Investigational Site, Bryanston
  - 1160.46.27013 Boehringer Ingelheim Investigational Site, Cape Town
  - 1160.46.27007 Boehringer Ingelheim Investigational Site, Centurion
  - 1160.46.27014 Boehringer Ingelheim Investigational Site, Kempton Park
  - 1160.46.27015 Boehringer Ingelheim Investigational Site, Krugersdorp
  - 1160.46.27002 Boehringer Ingelheim Investigational Site, Morningside
  - 1160.46.27012 Boehringer Ingelheim Investigational Site, Plumstead
  - 1160.46.27006 Boehringer Ingelheim Investigational Site, Sunninghill
- South Korea (9):
  - 1160.46.82007 Boehringer Ingelheim Investigational Site, Busan
  - 1160.46.82003 Boehringer Ingelheim Investigational Site, Goyang-si
  - 1160.46.82008 Boehringer Ingelheim Investigational Site, Gyeonggi-do
  - 1160.46.82010 Boehringer Ingelheim Investigational Site, Gyeonggi-do
  - 1160.46.82002 Boehringer Ingelheim Investigational Site, Kyunggi-do
  - 1160.46.82004 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.46.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.46.82006 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.46.82009 Boehringer Ingelheim Investigational Site, Seoul
- Spain (6):
  - 1160.46.34002 Boehringer Ingelheim Investigational Site, Barcelona
  - 1160.46.34007 Boehringer Ingelheim Investigational Site, Cartagena. Murcia
  - 1160.46.34009 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.46.34015 Boehringer Ingelheim Investigational Site, Palma de Mallorca
  - 1160.46.34014 Boehringer Ingelheim Investigational Site, Sabadell - Barcelona
  - 1160.46.34011 Boehringer Ingelheim Investigational Site, Valencia
- Sweden (5):
  - 1160.46.46002 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1160.46.46010 Boehringer Ingelheim Investigational Site, Kristianstad
  - 1160.46.46001 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.46.46008 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.46.46003 Boehringer Ingelheim Investigational Site, Uppsala
- Taiwan (5):
  - 1160.46.88607 Boehringer Ingelheim Investigational Site, Changhua
  - 1160.46.88604 Boehringer Ingelheim Investigational Site, Taipei
  - 1160.46.88606 Boehringer Ingelheim Investigational Site, Taipei
  - 1160.46.88608 Boehringer Ingelheim Investigational Site, Taipei
  - 1160.46.88609 Boehringer Ingelheim Investigational Site, Taipei
- Thailand (7):
  - 1160.46.66007 Boehringer Ingelheim Investigational Site, Bangkok
  - 1160.46.66010 Boehringer Ingelheim Investigational Site, Bangkok
  - 1160.46.66001 Boehringer Ingelheim Investigational Site, Khon Kaen
  - 1160.46.66004 Boehringer Ingelheim Investigational Site, Muang Nakhonratchasima
  - 1160.46.66005 Boehringer Ingelheim Investigational Site, Nakhonratchasima
  - 1160.46.66006 Boehringer Ingelheim Investigational Site, Nokorn Nayok
  - 1160.46.66008 Boehringer Ingelheim Investigational Site, Phayathai
- Turkey (Türkiye) (8):
  - 1160.46.90003 Boehringer Ingelheim Investigational Site, Ankara
  - 1160.46.90004 Boehringer Ingelheim Investigational Site, Ankara
  - 1160.46.90001 Boehringer Ingelheim Investigational Site, Istanbul
  - 1160.46.90002 Boehringer Ingelheim Investigational Site, Istanbul
  - 1160.46.90007 Boehringer Ingelheim Investigational Site, Istanbul
  - 1160.46.90008 Boehringer Ingelheim Investigational Site, Istanbul
  - 1160.46.90009 Boehringer Ingelheim Investigational Site, Istanbul
  - 1160.46.90010 Boehringer Ingelheim Investigational Site, Istanbul
- 1160.46.38005 Boehringer Ingelheim Investigational Site, Vinnitsa, Ukraine
- United Kingdom (5):
  - 1160.46.44005 Boehringer Ingelheim Investigational Site, Headington, Oxford
  - 1160.46.44011 Boehringer Ingelheim Investigational Site, London
  - 1160.46.44006 Boehringer Ingelheim Investigational Site, Newcastle upon Tyne
  - 1160.46.44013 Boehringer Ingelheim Investigational Site, Plymouth
  - 1160.46.44012 Boehringer Ingelheim Investigational Site, Sheffield

REFERENCES:
- [Derived] Goldhaber SZ, Eriksson H, Kakkar A, Schellong S, Feuring M, Fraessdorf M, Kreuzer J, Schueler E, Schulman S. Efficacy of dabigatran versus warfarin in patients with acute venous thromboembolism in the presence of thrombophilia: Findings from RE-COVER(R), RE-COVER II, and RE-MEDY. Vasc Med. 2016 Dec;21(6):506-514. doi: 10.1177/1358863X16668588. Epub 2016 Nov 1. PMID 27807306
- [Derived] Schulman S, Kakkar AK, Goldhaber SZ, Schellong S, Eriksson H, Mismetti P, Christiansen AV, Friedman J, Le Maulf F, Peter N, Kearon C; RE-COVER II Trial Investigators. Treatment of acute venous thromboembolism with dabigatran or warfarin and pooled analysis. Circulation. 2014 Feb 18;129(7):764-72. doi: 10.1161/CIRCULATIONAHA.113.004450. Epub 2013 Dec 16. PMID 24344086
- [Derived] Majeed A, Hwang HG, Connolly SJ, Eikelboom JW, Ezekowitz MD, Wallentin L, Brueckmann M, Fraessdorf M, Yusuf S, Schulman S. Management and outcomes of major bleeding during treatment with dabigatran or warfarin. Circulation. 2013 Nov 19;128(21):2325-32. doi: 10.1161/CIRCULATIONAHA.113.002332. Epub 2013 Sep 30. PMID 24081972

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 2589 patients enrolled/randomised but only 2568 were treated.
Groups:
- Dabigatran 150 mg: bid (twice daily) oral
- Warfarin: PRN (as needed) to maintain an INR (international normalised ratio) of 2.0-3.0
Period: Overall Study
Arm/Group | Dabigatran 150 mg | Warfarin
Started | 1280 (Started treatment.) | 1288 (Started treatment.)
Completed | 1155 (Completed planned observation time.) | 1172 (Completed planned observation time.)
Not Completed | 125 | 116
Not completed — Adverse Event | 47 | 44
Not completed — Protocol Violation | 31 | 26
Not completed — Lost to Follow-up | 11 | 6
Not completed — Withdrawal by Subject | 32 | 39
Not completed — Other | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Dabigatran 150 mg: bid oral
- Warfarin: PRN to maintain an INR of 2.0-3.0
- Total: Total of all reporting groups
Arm/Group | Dabigatran 150 mg | Warfarin | Total
Number analyzed (Participants) | 1280 | 1288 | 2568
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.7 (16.19) | 55.1 (16.26) | 54.9 (16.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 499 | 512 | 1011
  Male | 781 | 776 | 1557
Investigator assessed acute symptomatic deep vein thrombosis (DVT) of leg or pulmonary embolism (PE) [Number; unit: participants]
  Symptomatic PE and symptomatic DVT | 104 | 117 | 221
  Symptomatic PE | 298 | 297 | 595
  Symptomatic DVT | 877 | 873 | 1750
  No PE and no DVT | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrent Symptomatic Venous Thromboembolism (VTE) and Deaths Related to VTE
Description: All suspected recurrent VTEs and all deaths and bleeding events were evaluated by an independent central adjudication committee, and all analyses are based on the events that were centrally confirmed by this committee.
Time Frame: For statistical analysis 1: from randomisation to end of post treatment period (ptp), planned to be up to day 224. For statistical analysis 2: from randomisation to 6 months (up to day 180)
Population: Full analysis set (FAS): consisted of all randomised patients who were documented to have taken at least one dose of study drug. Patients were assigned to the treatment groups as randomised, i.e. regardless of the actual medication taken.
Measure: Number; unit: participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1279 | 1289
participants
  Participants with event (up to day 180) | 30 | 28
  Participants with event (up to end of ptp) | 34 | 30
Statistical Analysis 1: Comparison: Dabigatran 150 mg vs Warfarin; Hazard ratio (HR) vs. Warfarin (events occurring between randomisation and end of ptp). The time to first occurrence of the primary endpoint was compared between treatment groups using the Cox proportional hazards (PH) model, including the factors treatment, active cancer at baseline, symptomatic PE at baseline, and the interaction between active cancer and symptomatic PE; Test type: Non-Inferiority or Equivalence — Non inferiority margin was set up to 2.75 for the HR analysis; p = 0.0002, Regression, Cox — Non-inferiority P-Value.Two co-primary analyses performed on primary endpoint. Both non inferiority for the risk difference (RD) (at day 180) and for the HR (up to end of ptp) analyses to be reached in order to conclude positively on primary endpoint; Patients without events are censored at the end of ptp; Hazard Ratio (HR) = 1.13, 95% CI [0.69 to 1.85]
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; RD vs. Warfarin for Proportion of patients with VTE or death related to VTE at 6 months. Point estimate and 95% CI for the overall RD obtained based on the Kaplan Meier (KM) estimates at 6 months (180 days) after adjusting for the stratification factors active cancer at baseline and symptomatic PE at baseline; Test type: Non-Inferiority or Equivalence — Non inferiority margin was set up to 3.6% for the RD based on KM estimates; p < 0.0001, Kaplan Meier weighted estimates — Non-inferiority P-Value.Two co-primary analyses performed on primary endpoint. Both non inferiority for the RD (at day 180) and for the HR (events up to end of ptp) analyses to be reached in order to conclude positively on the primary endpoint; Risk Difference (Percentage) = 0.2, 95% CI [-1.0 to 1.3]
Statistical Analysis 3: Comparison: Dabigatran 150 mg vs Warfarin; HR vs. Warfarin (events occurring between randomisation and day 180). The time to first occurrence of the primary endpoint was compared between treatment groups using the Cox PH model, including the factors treatment, active cancer at baseline, symptomatic PE at baseline, and the interaction between active cancer and symptomatic PE. This analysis was performed as sensitivity analysis for statistical analysis 1; Test type: Superiority or Other; Regression, Cox; Patients without events are censored at the earliest of last contact date or day 180; Hazard Ratio (HR) = 1.08, 95% CI [0.64 to 1.8]

2. Secondary Outcome: Number of Participants With Recurrent Symptomatic VTE and All Deaths
Description: VTE or any death which occured from randomisation to end of ptp. All suspected recurrent VTEs and all deaths and bleeding events were evaluated by an independent central adjudication committee, and all analyses are based on the events that were centrally confirmed by this committee.
Time Frame: For statistical analysis 1: from randomisation to 6 months (up to day 180) For statistical analysis 2: from randomisation to end of ptp, planned to be up to day 224.
Population: FAS
Measure: Number; unit: participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1279 | 1289
participants
  Participants with event (up to day 180) | 51 | 48
  Participants with event (up to end of ptp) | 57 | 51
Statistical Analysis 1: Comparison: Dabigatran 150 mg vs Warfarin; RD vs. Warfarin for Proportion of patients with VTE or death at 6 months. Point estimate and 95% CI for the overall RD obtained based on the KM estimates at 6 months (180 days) after adjusting for the stratification factors active cancer at baseline and symptomatic PE at baseline; Test type: Superiority or Other; p = 0.6932, Kaplan Meier weighted estimates; Risk Difference (Percentage) = 0.3, 95% CI [-1.1 to 1.6]
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; HR vs. Warfarin (events occurring between randomisation and end of ptp). The time to first occurrence of the endpoint was compared between treatment groups using the Cox PH model, including the factors treatment, active cancer at baseline, symptomatic PE at baseline, and the interaction between active cancer and symptomatic PE; Test type: Superiority or Other; p = 0.6383, Regression, Cox; Patients without events are censored at the end of ptp; Hazard Ratio (HR) = 1.09, 95% CI [0.75 to 1.60]

3. Secondary Outcome: Number of Participants With Recurrent Symptomatic DVT
Description: Symptomatic DVT which occured from randomisation to end of ptp. All suspected recurrent VTEs and all deaths and bleeding events were evaluated by an independent central adjudication committee, and all analyses are based on the events that were centrally confirmed by this committee.
Time Frame: as for outcome 2
Population: FAS
Measure: Number; unit: participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1279 | 1289
participants
  Participants with event (up to day 180) | 25 | 17
  Participants with event (up to end of ptp) | 28 | 17
Statistical Analysis 1: Comparison: Dabigatran 150 mg vs Warfarin; RD vs. Warfarin for Proportion of patients with symptomatic DVT at 6 months. Point estimate and 95% CI for the overall RD obtained based on the KM estimates at 6 months (180 days) after adjusting for the stratification factors active cancer at baseline and symptomatic PE at baseline; Test type: Superiority or Other; p = 0.1703, Kaplan Meier weighted estimates; Risk Difference (Percentage) = 0.6, 95% CI [-0.3 to 1.5]
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.1054, Regression, Cox; Patients without events are censored at the end of ptp; Hazard Ratio (HR) = 1.65, 95% CI [0.90 to 3.01]

4. Secondary Outcome: Number of Participants With Recurrent Symptomatic Non-fatal PE
Description: Symptomatic non-fatal PE which occured from randomisation to end of ptp. All suspected recurrent VTEs and all deaths and bleeding events were evaluated by an independent central adjudication committee, and all analyses are based on the events that were centrally confirmed by this committee.
Time Frame: For statistical analysis 1: from randomisation to 6 months (up to day 180). For statistical analysis 2: from randomisation to end of ptp, planned to be up to day 224.
Population: FAS
Measure: Number; unit: participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1279 | 1289
participants
  Participants with event (up to day 180) | 7 | 13
  Participants with event (up to end of ptp) | 9 | 15
Statistical Analysis 1: Comparison: Dabigatran 150 mg vs Warfarin; RD vs. Warfarin for Proportion of patients with symptomatic non-fatal PE at 6 months. Point estimate and 95% CI for the overall RD obtained based on the KM estimates at 6 months (180 days) after adjusting for the stratification factors active cancer at baseline and symptomatic PE at baseline; Test type: Superiority or Other; p = 0.2283, Kaplan Meier weighted estimates; Risk Difference (Percentage) = -0.4, 95% CI [-1.1 to 0.3]
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.2101, Regression, Cox; Hazard Ratio (HR) = 0.59, 95% CI [0.26 to 1.35]

5. Secondary Outcome: Number of Participants Who Died Due to VTE
Description: VTE - related deaths which occured from randomisation to end of ptp. All suspected recurrent VTEs and all deaths and bleeding events were evaluated by an independent central adjudication committee, and all analyses are based on the events that were centrally confirmed by this committee. Hazard ratios and 95% CI were not calculated because of insufficient number of events.
Time Frame: From randomisation to 6 months (up to day 180) and to end of ptp (planned to be up to day 224)
Population: FAS
Measure: Number; unit: participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1279 | 1289
participants
  Participants with event (up to day 180) | 3 | 0
  Participants with event (up to end of ptp) | 3 | 0
Statistical Analysis 1: Comparison: Dabigatran 150 mg vs Warfarin; RD at 6 months vs. Warfarin for Proportion of patients who died due to VTE . Point estimate and 95% CI for the overall RD obtained based on the KM estimates at 6 months (180 days) after adjusting for the stratification factors active cancer at baseline and symptomatic PE at baseline; Test type: Superiority or Other; p = 0.0830, Kaplan Meier weighted estimates; Risk Difference (Percentage) = 0.2, 95% CI [0.0 to 0.5]

6. Secondary Outcome: Number of Participants Who Died (Any Cause)
Description: Any deaths which occured from randomisation to end of ptp. All suspected recurrent VTEs and all deaths and bleeding events were evaluated by an independent central adjudication committee, and all analyses are based on the events that were centrally confirmed by this committee.
Time Frame: as for outcome 2
Population: FAS
Measure: Number; unit: participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1279 | 1289
participants
  Participants with event (up to day 180) | 25 | 25
  Participants with event (up to end of ptp) | 29 | 26
Statistical Analysis 1: Comparison: Dabigatran 150 mg vs Warfarin; RD at 6 months vs. Warfarin for Proportion of patients who died from any cause. Point estimate and 95% CI for the overall RD obtained based on the KM estimates at 6 months (180 days) after adjusting for the stratification factors active cancer at baseline and symptomatic PE at baseline; Test type: Superiority or Other; p = 0.7348, Kaplan Meier weighted estimates; Risk Difference (Percentage) = 0.1, 95% CI [-0.7 to 1.0]
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.8939, Regression, Cox; Patients without events are censored at the end of ptp; Hazard Ratio (HR) = 1.04, 95% CI [0.61 to 1.77]

7. Secondary Outcome: Number of Participants With Recurrent Symptomatic Fatal and Non-fatal PE
Description: Symptomatic fatal and non-fatal PE which occured from randomisation to end of ptp. All suspected recurrent VTEs and all deaths and bleeding events were evaluated by an independent central adjudication committee, and all analyses are based on the events that were centrally confirmed by this committee.
Time Frame: as for outcome 4
Population: FAS
Measure: Number; unit: participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1279 | 1289
participants
  Participants with event (up to day 180) | 8 | 13
  Participants with event (up to end of ptp) | 10 | 15
Statistical Analysis 1: Comparison: Dabigatran 150 mg vs Warfarin; RD vs. Warfarin for Proportion of patients with symptomatic fatal and non-fatal PE at 6 months. Point estimate and 95% CI for the overall RD obtained based on the KM estimates at 6 months (180 days) after adjusting for the stratification factors active cancer at baseline and symptomatic PE at baseline; Test type: Superiority or Other; p = 0.3210, Kaplan Meier weighted estimates; Risk Difference (Percentage) = -0.3, 95% CI 2-sided [-1.0 to 0.3]
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.3021, Regression, Cox; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.29 to 1.46]

8. Secondary Outcome: Number of Participants With MBE, MBE and/or CRBE, and Any Bleeding Events
Description: Major bleeding events (MBE) are defined as
  * Fatal bleeding
  * Symptomatic bleeding in a critical area or organ
  * Bleeding causing a fall in haemoglobin level of 20 g/L (1.24 mmol/L) or more, or leading to transfusion of 2 or more units of whole blood or red cells
  Clinically-relevant bleeding events (CRBE) are defined as
  * spontaneous skin hematoma >=25 cm²
  * wound hematoma >=100 cm²
  * spontaneous nose bleed >5 min
  * macroscopic hematuria spontaneous or >24 hours if associated with an intervention
  * spontaneous rectal bleeding
  * gingival bleeding >5 min
  * leading to hospitalisation and / or requiring surgical treatment
  * leading to a transfusion of <2 units of whole blood or red cells
  * any other bleeding event considered clinically relevant by the investigator
  Any bleeding events were defined as major, clinically-relevant and nuisance bleeding events. Nuisance bleeding events were defined as all other bleeding events that did not fulfil the criteria from above.
Time Frame: From first intake of study drug to last intake of study drug + 6 days washout
Population: Treated set (TS): consisted of all randomised patients who were documented to have taken at least one dose of study drug. Patients were assigned to the treatment groups as treated.
Measure: Number; unit: participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1280 | 1288
participants
  MBE | 15 | 22
  MBE and/or CRBE | 64 | 102
  Any bleeding event | 200 | 285
Statistical Analysis 1: Comparison: Dabigatran 150 mg vs Warfarin; HR vs. Warfarin (events occurring between 1st intake of study drug and last intake of study drug + 6 days). The time to first occurrence of MBE was compared between treatment groups using the Cox PH model, including the factors treatment, active cancer at baseline, symptomatic PE at baseline, and the interaction between active cancer and symptomatic PE; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 0.69, 95% CI [0.36 to 1.32] — This is the analysis of the time to the first MBE
Statistical Analysis 2: Comparison: Dabigatran 150 mg vs Warfarin; HR vs. Warfarin (events occurring between 1st intake of study drug and last intake of study drug + 6 days). The time to first occurrence of any bleeding was compared between treatment groups using the Cox PH model, including the factors treatment, active cancer at baseline, symptomatic PE at baseline, and the interaction between active cancer and symptomatic PE; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.56 to 0.81] — This is the analysis of the time to the first occurrence of any bleeding event

9. Secondary Outcome: Number of Participants With Acute Coronary Syndrome (ACS)
Description: Any ACS occurring during the conduct of the study (centrally adjudicated as definite). Patients having a centrally adjudicated definite ACS during intake of study drug and after stopping study drug, according to treatment group. ACS assessments pre-specified in the protocol without adjudication. Prior to database lock, the steering committee asked to have ACS events adjudicated by an independent committee. After database lock, the committee was provided with source documentation that was blinded to the patient's treatment assignment. ACS results presented are based on adjudication findings.
Time Frame: From first intake of study drug to last contact date
Population: TS
Measure: Number; unit: participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1280 | 1288
participants
  During intake of study drug | 3 | 0
  After stopping study drug | 2 | 1

10. Secondary Outcome: Laboratory Analyses
Description: Frequency of patients with possible clinically significant abnormalities.
Time Frame: From first intake of study drug to last intake of study drug + 6 days washout
Population: TS
Measure: Number; unit: participants
Arm/Group | Dabigatran 150 mg | Warfarin
Number analyzed (Participants) | 1238 | 1248
participants
  AST increase | 29 | 27
  AST decrease | 0 | 0
  ALT increase | 31 | 40
  ALT decrease | 0 | 0
  Bilirubin increase | 8 | 6
  Bilirubin decrease | 0 | 0

ADVERSE EVENTS:
Time Frame: From first intake of study drug to last intake of study drug + 6 days washout
Arm/Group | Dabigatran 150 mg | Warfarin
Serious Adverse Events (participants affected / at risk) | 156/1280 | 153/1288
Other Adverse Events (participants affected / at risk) | 124/1280 | 126/1288
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran 150 mg (N=1280) | Warfarin (N=1288)
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 2
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 4 | 0
Angina unstable (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 3 | 0
Cardiac failure (Cardiac disorders) | 1 | 3
Cardiac failure congestive (Cardiac disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 1
Caecitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastritis alcoholic (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1
Ileal fistula (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 1 | 1
Chest pain (General disorders) | 7 | 5
Death (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 2
Pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Behcet's syndrome (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 2
Abdominal abscess (Infections and infestations) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 1
Bone abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 5 | 4
Erysipelas (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 9 | 4
Pulmonary tuberculoma (Infections and infestations) | 1 | 0
Purulent pericarditis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 3 | 4
Subcutaneous abscess (Infections and infestations) | 0 | 1
Syphilis (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 4
Urosepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Incision site haematoma (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Radial nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Snake bite (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Coagulation time prolonged (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 1 | 1
International normalised ratio fluctuation (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 2
Prothrombin time prolonged (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteodystrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pseudomyxoma peritonei (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 2
Haematuria (Renal and urinary disorders) | 3 | 9
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 2
Renal impairment (Renal and urinary disorders) | 0 | 1
Renal vein thrombosis (Renal and urinary disorders) | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Pelvic haematoma (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 14 | 9
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Social problem (Social circumstances) | 1 | 0
Intestinal operation (Surgical and medical procedures) | 1 | 0
Tenotomy (Surgical and medical procedures) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 13 | 8
Embolism venous (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 1
Haemorrhage (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 1
Vascular compression (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran 150 mg (N=1280) | Warfarin (N=1288)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 75 | 69
Headache (Nervous system disorders) | 57 | 70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.